CLINICAL TRIAL: NCT00915252
Title: A Randomized, Multi-center Phase II Trial to Assess the Efficacy of 5-azacytidine Added to Standard Primary Therapy in Elderly Patients With Newly Diagnosed AML
Brief Title: Efficacy of 5-azacytidine Added to Standard Primary Therapy in Elderly Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Acronym: AML-AZA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Celgene Corporation (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101010
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; azacitidine; elderly; demethylating agent; flt3; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-azacytidine (Experimental): Patients enrolled in this arm will receive standard induction and consolidation chemotherapy preceded by 5-azacytidine. These patients will additionally receive maintenance therapy with 5-azacytidine for one year after start of induction therapy.
  Interventions: Drug: azacitidine
- standard chemotherapy (Active Comparator): Patients enrolled in this arm will receive standard chemotherapy treatment.
  Interventions: Drug: standard chemotherapy (7+3 scheme): Daunorubicin, Cytarabine

INTERVENTIONS:
Drug: azacitidine — Starting dose has been determined during run-in dose finding part of the study. Starting dose of the interventional drug is 75 mg/m²/d. Application form:
  During induction therapy phase: i.v. on days -5--1 before standard chemotherapy for 1 or 2 cycles, During consolidation therapy: s.c. on days -5--1 before standard chemotherapy (2 cycles).
  During maintenance therapy: s.c. on days 1-5 on a 28day cycle till maximum one year after start of first induction therapy.
  Other Names: 5-azacytidine; Vidaza
  Arms: 5-azacytidine
Drug: standard chemotherapy (7+3 scheme): Daunorubicin, Cytarabine — Induction therapy:
  Daunorubicin 60mg/m²/d i.v.on days 3,4,5 AraC 100mg/m²/d i.v. on days 1-7
  Consolidation therapy:
  AraC 1g/m² twice a day on day 1,3,5
  Other Names: Ara-C; Daunoblastin; DaunoXome; Alexan; Ara-cell; Udicil
  Arms: standard chemotherapy

SUMMARY:
The primary purpose of the study is to determine, whether the addition of 5-azacytidine to standard chemotherapy in elderly patients with newly diagnosed AML improves treatment results (event free survival).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML (except APL) according to the FAB or WHO classification, including AML evolving from MDS or other hematological diseases and AML after previous cytotoxic therapy or radiation (secondary AML).
* Bone marrow aspirate or biopsy must contain ≥ 20% blasts of all nucleated cells or differential blood count must contain ≥ 20% blasts. In AML FAB M6 ≥ 30% of non-erythroid cells in the bone marrow must be leukemic blasts. In AML defined by cytogenetic aberrations the proportion of blasts may be < 20%.
* Age ≥ 61 years
* Informed consent, personally signed and dated to participate in the study
* Male patients enrolled in this trial must use adequate barrier birth control measures during the course of the 5-azacytidine treatment and for at least 3 months after the last administration of 5-azacytidine.

Exclusion Criteria:

* Patients who are not eligible for standard chemotherapy as described in chapter 5.2 and 5.3
* Hyperleukocytosis (leukocytes > 20,000/µl) at study entry. These patients should be treated with hydroxyurea or receive leukocytapheresis treatment (if leukocytes > 100,000/µl) according to routine practice and entered into the study when leukocyte counts below 20,000/µl are reached. This applies only for the controlled part of the study.
* Patients with initial hyperleukocytosis above 20,000/µl can only be enrolled into the controlled part of the study, but not in the run-in dose finding part.
* Known central nervous system manifestation of AML
* Cardiac Disease: Heart failure NYHA class 3 or 4; unstable coronary artery disease (MI more than 6 months prior to study entry is permitted); serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Chronically impaired renal function (creatinin clearance < 30 ml / min)
* Inadequate liver function (ALT and AST ≥ 2.5 x ULN) if not caused by leukemic infiltration
* Total bilirubin ≥ 1.5 x ULN if not caused by leukemic infiltration
* Known HIV and/or hepatitis C infection
* Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy
* Evidence or recent history of CNS disease, including primary or metastatic brain tumors, seizure disorders
* Uncontrolled active infection
* Concurrent malignancies other than AML with an estimated life expectancy of less than two years
* History of organ allograft
* Hypersensitivity to cytarabine (not including drug fever or exanthema), daunorubicin, azacytidine or mannitol
* Previous treatment of AML except hydroxyurea and up to 2 days of ≤100 mg/m2/d cytarabine
* Previous therapy with 5-azacytidine (i.e. for an antecedent myelodysplastic syndrome)
* Patients with investigational drug therapy outside of this trial during or within 4 weeks of study entry should be discussed with the study office whether study participation is possible
* Any severe concomitant condition, which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Median Event Free Survival (EFS) of all AML patients | continously up to 12 months after start of study

SECONDARY OUTCOMES:
Median event free survival of AML patients with different cytogenetic and molecular risk groups | continously up to 12 months after study start
Median overall survival of all AML patients | continously up to 12 month after start of study
Median overall survival of AML patients with different cytogenetic and molecular risk groups | continously up to 12 month after start of study
Relapse free survival | continously up to 12 months after start of study

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Müller-Tidow, MD, Principal Investigator — Universitätsklinikum Münster, Medizinische Klinik A
Locations (27):
- Germany (27):
  - RWTH Aachen, Medizinische Klinik IV, Aachen
  - Sozialstiftung Bamberg, Klinikum am Bruderwald, Med. Klinik V, Bamberg
  - Klinikum Bayreuth, Medizinische Klinik IV, Bayreuth
  - Charite Campus Benjamin Franklin, Universitätsmedizin Berlin, Medizinische Klinik III, Berlin
  - Städt. Kliniken Bielefeld gem. GmbH, Klinikum Mitte, Klinik für Hämatologie, Onkologie, Palliativmedizin, Bielefeld
  - Klinikum Chemnitz, Krankenhaus Küchenwald, Klinik für Innere Medizin III, Chemnitz
  - Universitätsklinikum Carl Gustav Carus, Medizinische Klinik und Poliklinik I, Dresden
  - Katholische Krankenhaus Duisburg, Duisburg
  - Universitätsklinikum Erlangen, Medizinische Klinik 5, Erlangen
  - Universitätsklinikum Essen, Klinik für Hämatologie, Essen
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Klinikum der Johann Wolfgang Goethe-Universität Frakfurt am Main, Frankfurt am Main
  - Asklepios Klinik St. Georg, Hämatologische Abteilung, Hamburg
  - St. Bernward Krankenhaus Hildesheim, Medizinische Klinik II, Hildesheim
  - Westpfalz-Klinikum GmbH, Med. Klinik I, Kaiserslautern
  - Stiftungsklinikum Mittelrhein, Hämatologie/ Onkologie, Koblenz
  - Johannes Gutenberg-Universität Mainz Klinikum, III. Medizinische Klinik und Poliklinik, Mainz
  - Phillips Universität Marburg, Fachbereich 20, ZIM, Marburg
  - Klinikum rechts der Isar, III. Medizinische Klinik, München
  - Universitätsklinikum Münster, Medizinische Klinik und Poliklinik A, Münster
  - Klinikum Nürnberg, Medizinische Klinik 5, Nuremberg
  - Klinikum Osnabrück, Klinik für Onkologie, Hämatologie, Immunologie, Osnabrück
  - Klinikum der Universität Regensburg, Klinik und Poliklinik für Innere Medizin I, Regensburg
  - Robert-Bosch-Krankenhaus, Zentrum für Innere Medizin, Stuttgart
  - Klinikum Mutterhaus der Borromäerinnen, Innere Medizin I, Trier
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik II, Würzburg

REFERENCES:
- [Derived] Krug U, Koschmieder A, Schwammbach D, Gerss J, Tidow N, Steffen B, Bug G, Brandts CH, Schaich M, Rollig C, Thiede C, Noppeney R, Stelljes M, Buchner T, Koschmieder S, Duhrsen U, Serve H, Ehninger G, Berdel WE, Muller-Tidow C. Feasibility of azacitidine added to standard chemotherapy in older patients with acute myeloid leukemia--a randomised SAL pilot study. PLoS One. 2012;7(12):e52695. doi: 10.1371/journal.pone.0052695. Epub 2012 Dec 31. PMID 23300745